CLINICAL TRIAL: NCT05462301
Title: Normal Reference Range for Neonatal Echocardiography: a Multi-center, Prospective Study
Brief Title: Normal Reference Range for Neonatal Echocardiography
Acronym: NORRNE
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Collaborators: Shanxi Provincial Maternity and Children's Hospital (Other); Inner Mongolia Maternal and Child Health Care Hospital (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Ningxia Medical University (Other)
Responsible Party: Principal Investigator, Wang Jianhui, Project Leader, Children's Hospital of Chongqing Medical University
Other Study IDs: 2022-06-10
Record Dates: First submitted 2022-06-25; First posted 2022-07-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Echocardiography
Keywords: Neonatal Echocardiogram; Reference Ranges; Preterm Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — Neonatal bedside echocardiography was performed by a trained neonatologist or sonographer

SUMMARY:
Echocardiography is the main method of bedside examination of neonatal cardiac morphology, which can timely diagnose congenital heart disease and quantitatively assess its severity, but the diagnosis and evaluation process depends on the normal range of neonatal echocardiography.At present, there have been normal reference standards for echocardiography in children and adults at home and abroad, but there is no uniform standard for echocardiographic parameters in newborns, especially premature infants.This study intends to carry out a national multicenter, prospective, observational study to establish the reference range of echocardiography at different time periods after birth in newborns, and stratified according to gestational age, birth weight and gender, to conduct a more accurate hemodynamic assessment of clinically critically ill newborns and guide the treatment of critically ill newborns in real time.

DETAILED DESCRIPTION:
Neonatal goal-directed echocardiography (TNE) performed by neonatologists has been increasingly applied to hemodynamic assessment in the NICU to guide critical neonatal treatment in real time. There are many detection indexes of TNE, which are closely related to neonatal weight, birth weight, postnatal age, race and other factors. Therefore, establishing neonatal echocardiographic reference ranges is essential for the development of TNE. At present, there have been normal reference standards for echocardiography in children and adults at home and abroad, but there is no uniform standard for echocardiographic parameters in newborns, especially premature infants. At present, there are many problems in establishing the reference range of neonatal echocardiography internationally, including the small sample size included in establishing the reference range, no premature infant standard for some parameters, the reference range is not stratified according to gender, etc. Moreover, the majority of current echocardiographic reference ranges are derived from studies in European and American populations and are not applicable to Asian patients. So far, reference ranges for neonatal echocardiography established based on high-quality clinical studies are still lacking, greatly affecting the use of echocardiography in neonatal intensive care units. Therefore, this study intends to carry out a national multicenter, prospective, observational study to establish the reference range of echocardiography at different time periods after birth in neonates, and stratify according to creatinine, birth weight and gender, providing a reference for the application of echocardiography in neonatal intensive care units, and providing an important basis for the development of TNE-centered neonatal hemodynamic comprehensive assessment program in the NICU.

1. Study Design and Process:

   This study is a multicenter, prospective, observational study. Neonatal bedside echocardiography was performed by a trained neonatology clinician or sonographer. Five time points were selected for neonatal echocardiography, namely, 1 day, 3 days, 7 days, 14 days, and 28 days after birth. The examination was completed in the quiet state of the newborn, and the measurement method was based on the American Guidelines and Standards for Echocardiography in Children and the American NICU Echocardiography Practice Guidelines. All ultrasound data were averaged over three or more cardiac cycles.
2. Sample Size Calculation:

   Each participating NICU will be required to enroll 300 infants (60 infants for each PNA timepoint) for a final sample size of 1500 "normal infants".
3. Statistical Methods:

   Data statistics were performed using SPSS 21.0 software. The data obtained for each of the ultrasound hemodynamic parameters were tested for normality. The measurement data conforming to normal distribution are expressed by mean ± standard deviation, and the measurement data with non-normal distribution are expressed by median (interquartile range). Spearman correlation analysis was used to compare the correlation between different indicators and postnatal, birth weight, birth weight and gender. The echocardiographic reference range of newborns at different time periods after birth was established by 95% confidence interval and stratified according to birth weight, birth weight and gender. P < 0.05 was considered statistically significant.
4. Quality control:

At the beginning of the study, a cooperative group kick-off meeting will be organized to interpret the study protocol in detail. In addition, the online or offline training of the participating units will be carried out to further unify the parameter setting and data collection criteria of the ultrasound machine. Establish a WeChat group to answer questions related to this study at any time. During the process of the project, regular contact meetings within the cooperative group will be held to ensure that the investigators participating in the study will implement the protocol. During the study, the study site will assign a special person to review the completeness and correctness of the data submitted by each participating site.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient or inpatient neonate
* Gestational age > 30weeks and birthweight > 1250 grams
* Appropriate for gestational age
* Without perinatal asphyxia
* Without skin lesion on the left chest wall
* with family informed consent for neonatal echocardiography

Exclusion Criteria:

* specialist cardiac ultrasound suggests congenital heart disease;
* PDA with hemodynamic abnormalities, defined as: PDA > 1.5 mm (left-to-right shunt) and left atrial diameter/aortic root > 1.5 or the need for the use of inotropes;
* invasive mechanical ventilation therapy,
* non-invasive mechanical ventilation with FiO2 >0.3
* major anomalies
* blood culture-proven neonatal sepsis
* persistent pulmonary hypertension
* renal failure
* necrotizing enterocolitis ≥ stage II
* post surgery
* Maternal history of severe anemia, or prenatal massive bleeding

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy neonates and preterm Infants
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in left atrial anteroposterior diameter with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  The Left atrial systolic anteroposterior diameter was measured by M-mode ultrasound through the aortic root in the long axis of the parasternal left ventricle
Changes in interventricular septum thickness with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  The Interventricular septal thickness was measured by left ventricular M-mode ultrasound in the long axis of the parasternal left ventricle
Changes in left ventricular posterior wall thickness at end diastole with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  The left ventricular posterior wall thickness at end diastole was measured by left ventricular M-mode ultrasound in the long axis of the parasternal left ventricle
Changes in left ventricular end diastolic diameter with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  The left ventricular end diastolic diameter was measured by left ventricular M-mode ultrasound in the long axis of the parasternal left ventricle
Changes in left ventricular end systolic diameter with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  The left ventricular end systolic diameter was measured by left ventricular M-mode ultrasound in the long axis of the parasternal left ventricle
Changes in right ventricular anteroposterior diameter at end diastole with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  The right ventricular anteroposterior diameter at end diastole was measured by left ventricular M-mode ultrasound in the long axis of the parasternal left ventricle
Changes in right ventricular outflow tract diameter with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  The right ventricular outflow tract diameter was measured in the short-axis pulmonary valve orifice view of the parasternal great arteries
Changes in left ventricular ejection fraction with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  Left ventricular ejection fraction can be calculated by measuring left ventricular end-diastolic diameter and left ventricular end-systolic diameter in a standard parasternal left ventricular long-axis view, at the level of mitral chordae tendineae, or parasternal left ventricular short-axis view, at the level of papillary muscles, with the sampling line perpendicular to the interventricular septum and left ventricular posterior wall

SECONDARY OUTCOMES:
Changes in left ventricular outflow tract diameter with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  In the standard parasternal long-axis view, images were frozen when the aortic valve was completely opened during systole, and the distance between the anterior and posterior aortic walls at the level of aortic root attachment was measured with an electronic cursor to obtain the left ventricular outflow tract diameter
Changes in main pulmonary artery diameter with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  In the parasternal cardiac base short-axis view, the left and right pulmonary arteries were exposed at the same time, and the diameter of the main pulmonary artery was measured
Changes in Inferior vena cava diameter with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  Inferior vena cava diameter was measured by M-mode ultrasound in the subxiphoid long-axis plane by transthoracic ultrasound
Changes in Simpson 's method for measuring ejection fraction with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  Through the apical four-chamber view or apical two-chamber view, for the tracing of diastolic and systolic endocardium, divide the heart into several (generally 20) cylinders, calculate the volume and add them to obtain the left ventricular end-diastolic and end-systolic volumes, and then calculate the ejection fraction

OTHER OUTCOMES:
Changes in Aortic Velocity Time Integral（VTI）with increasing age | 5 time points (1 day, 3 days, 7 days, 14 days and 28 days after birth)
  In the apical five-chamber view, select the color Doppler mode to display the aortic blood flow signal and direction, place the sampling volume below the arterial orifice, adjust the blood flow direction as parallel as possible to the sampling line through the left and right swing probe, and select the pulsed Doppler mode (PW), then the velocity time integral (VTI) image of aortic blood flow can be obtained. Trace the aortic velocity-time integral image and calculate the VTI value in cm by computer or plotter. Select 3-5 consecutive VTI images within the same respiratory cycle for measurement and average to reduce the impact of the respiratory cycle

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jianhui, Doctor, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El-Khuffash A, Herbozo C, Jain A, Lapointe A, McNamara PJ. Targeted neonatal echocardiography (TnECHO) service in a Canadian neonatal intensive care unit: a 4-year experience. J Perinatol. 2013 Sep;33(9):687-90. doi: 10.1038/jp.2013.42. Epub 2013 Apr 25. PMID 23619373
- [Result] Shiraishi H, Yanagisawa M. Pulsed Doppler echocardiographic evaluation of neonatal circulatory changes. Br Heart J. 1987 Feb;57(2):161-7. doi: 10.1136/hrt.57.2.161. PMID 3814451
- [Result] Kluckow M, Evans N. Superior vena cava flow in newborn infants: a novel marker of systemic blood flow. Arch Dis Child Fetal Neonatal Ed. 2000 May;82(3):F182-7. doi: 10.1136/fn.82.3.f182. PMID 10794783
- [Result] Schmitz L, Stiller B, Pees C, Koch H, Xanthopoulos A, Lange P. Doppler-derived parameters of diastolic left ventricular function in preterm infants with a birth weight <1500 g: reference values and differences to term infants. Early Hum Dev. 2004 Feb;76(2):101-14. doi: 10.1016/j.earlhumdev.2003.11.003. PMID 14757262
- [Result] Cosyns B, Lancellotti P. Normal reference values for echocardiography: a call for comparison between ethnicities. Eur Heart J Cardiovasc Imaging. 2016 May;17(5):523-4. doi: 10.1093/ehjci/jev353. Epub 2016 Mar 13. No abstract available. PMID 26976356